CLINICAL TRIAL: NCT00114244
Title: A Randomized Phase II Study of BAY 43-9006 in Combination With Gemcitabine in Metastatic Pancreatic Carcinoma
Brief Title: Sorafenib With or Without Gemcitabine in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02835; NCI-2012-02835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-50 (Other: City of Hope); 6576 (Other: CTEP); N01CM62209 (NIH)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2013-10

CONDITIONS: Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sorafenib; Gemcitabine

ARMS (2):
- Arm I (sorafenib tosylate) (Experimental): Patients receive 400 mg oral sorafenib twice daily on days 1-28. Patients experiencing disease progression cross over to Arm II.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis
- Arm II (sorafenib tosylate, gemcitabine hydrochloride) (Experimental): Patients receive 400 mg oral sorafenib as in Arm I and 1000 mg/m2 gemcitabine IV over 100 minutes on days 1, 8, and 15.
  Interventions: Drug: sorafenib tosylate; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
  Arms: Arm II (sorafenib tosylate, gemcitabine hydrochloride)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II is studying how well giving sorafenib with or without gemcitabine works in treating patients with metastatic pancreatic cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with gemcitabine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate in patients with metastatic pancreatic cancer treated with concurrent gemcitabine and BAY43-9006 and sequential BAY 43-9006 followed by gemcitabine/BAY 43-9006 at progression.

SECONDARY OBJECTIVES:

I. To determine the six month overall survival rate, 3 month progression free survival rate, time to tumor progression and overall survival of patients with metastatic pancreatic cancer treated with concurrent gemcitabine and BAY43-9006 and sequential BAY 43-9006 followed by gemcitabine/BAY 43-9006 at progression.

II. To determine the safety profile of gemcitabine and BAY43-9006 in patients with metastatic pancreatic cancer and compared to those treated with single agent BAY 43-9006.

III. To determine whether mRNA expression levels of genes involved in the gemcitabine pathway (RR, dck, dcd) and genes involved in the Raf pathway (cyclin D, VEGFR2, p21) will predict for time to progression, overall survival, and response, in patients with metastatic pancreatic cancer treated with concurrent gemcitabine and BAY43-9006 and sequential BAY 43-9006 followed by gemcitabine/BAY 43-9006 at progression.

IV. To determine whether genomic polymorphisms of genes (measured in peripheral blood mononuclear cells) involved in the gemcitabine pathway (RR) and genes involved in the ras pathway (VEGFR2, cyclin D, p21) will predict for time to progression, overall survival, tumor response, and toxicity in patients with advanced cancer of the pancreas treated with concurrent gemcitabine and BAY43-9006 and sequential BAY 43-9006 followed by gemcitabine/BAY 43-9006 at progression.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral sorafenib twice daily on days 1-28. Patients experiencing disease progression cross over to Arm II.

ARM II: Patients receive oral sorafenib as in Arm I and gemcitabine IV over 100 minutes on days 1, 8, and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic pancreatic carcinoma
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* No prior chemotherapy for metastatic disease is allowed; prior adjuvant chemotherapy is allowed provided that patients did not receive gemcitabine and the chemotherapy completed > 6 months prior to initiation of study therapy
* Available tumor biopsy specimen (paraffin embedded or fresh frozen) that was obtained at the time of diagnosis and/or prior to study entry is required
* Life expectancy of greater than 3 months
* ECOG performance status =< 1
* Leukocytes >= 3,000/μL
* Absolute neutrophil count >= 1,500/μL
* Platelets >= 100,000/μL
* Hemoglobin >= 9 mg/dL
* Total bilirubin =< 1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 3 X institutional upper limit of normal, unless the liver is involved with tumor, in which the AST (SGOT)/ALT (SGPT) must be =< 5 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2
* The effects of BAY 43-9006 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because raf kinase inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Because BAY 43-9006 is at least partially metabolized by the CYP 3A enzyme in the liver, the possible effect that inhibitors of CYP 3A may have on BAY 43-9006 is unknown; therefore, patients taking inhibitors of CYP 3A (such as ketoconazole, itraconazole, and ritonavir) may not be enrolled in this study
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006 or gemcitabine
* Secondary primary malignancy (except in situ carcinoma of the cervix, in situ cancer of the prostate, in situ cancer of the breast or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 5 years previously with no evidence of recurrence); concurrent or history of another malignancy =< 5 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because BAY 43-9006 is a kinase inhibitor agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 43-9006, breastfeeding should be discontinued if the mother is treated with BAY 43-9006
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BAY 43-9006; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients with evidence of bleeding diathesis
* Patients receiving therapeutic doses of anticoagulation; prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride)
Started | 15 | 37
Completed | 13 | 30
Not Completed | 2 | 7
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride) | Total
Number analyzed (Participants) | 15 | 37 | 52
Age, Continuous [Median (Full Range); unit: years] | 66 [55 to 82] | 65 [43 to 83] | 65 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 21
  Male | 9 | 22 | 31
Region of Enrollment [Number; unit: participants]
  United States | 15 | 37 | 52

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR = CR or PR) as Determined by the RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan, MRI, X-ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Every 6 weeks.
Measure: Number; unit: participants
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 15 | 37
participants | 0 | 1

2. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier by arm.
Time Frame: From first day of treatment to time of death due to any cause, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 15 | 37
Months | 4.3 [3.3 to 8.3] | 6.5 [5.5 to 8.0]

3. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier by arm. The probability of progression-free survival at 3 months and overall survival at 6 months, and their Greenwood's standard errors will be summarized by arm.
Time Frame: From first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 3 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 15 | 37
Months | 2.3 [1.2 to 5.7] | 2.9 [2.1 to 4.3]

ADVERSE EVENTS:
Time Frame: Adverse Events occured over a 36 month period.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride): Patients receive 400 mg oral sorafenib as in Arm I and gemcitabine IV over 100 minutes on days 1, 8, and 15.
  sorafenib tosylate: Given PO
  gemcitabine hydrochloride: Given IV
  laboratory biomarker analysis: Correlative studies
Arm/Group | Arm I (Sorafenib Tosylate) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 8/15 | 15/37
Other Adverse Events (participants affected / at risk) | 15/15 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sorafenib Tosylate) (N=15) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride) (N=37)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Hyperbilirubinemia (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Sorafenib Tosylate) (N=15) | Arm II (Sorafenib Tosylate, Gemcitabine Hydrochloride) (N=37)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (13) | 17 (49)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular flutter (Cardiac disorders) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 10 (17) | 21 (45)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 7 (9) | 14 (32)
Diarrhea (Gastrointestinal disorders) | 5 (18) | 16 (36)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 5 (6)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 4 (6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastro-intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (5)
Nausea (Gastrointestinal disorders) | 8 (13) | 14 (23)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (8) | 8 (10)
Chills (General disorders) | 0 (0) | 7 (7)
Death (General disorders) | 1 (1) | 7 (7)
Disease progression (General disorders) | 11 (11) | 18 (18)
Edema limbs (General disorders) | 1 (1) | 4 (8)
Fatigue (General disorders) | 10 (33) | 27 (64)
Fever (General disorders) | 1 (1) | 4 (4)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
General symptom (General disorders) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2)
Pericardial pain (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Alanine aminotransferase increased (Investigations) | 2 (3) | 19 (40)
Alkaline phosphatase increased (Investigations) | 5 (14) | 22 (41)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 18 (43)
Creatinine increased (Investigations) | 0 (0) | 1 (2)
Hyperbilirubinemia (Investigations) | 2 (3) | 6 (7)
Leukocyte count decreased (Investigations) | 0 (0) | 3 (3)
Leukopenia (Investigations) | 1 (6) | 9 (18)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Lymphopenia (Investigations) | 1 (3) | 7 (13)
Neutrophil count decreased (Investigations) | 2 (6) | 17 (29)
Platelet count decreased (Investigations) | 3 (10) | 21 (54)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (5) | 10 (15)
Anorexia (Metabolism and nutrition disorders) | 7 (17) | 21 (38)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (10) | 14 (29)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (6) | 8 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (5) | 9 (16)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 8 (16)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 6 (8)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 5 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (7)
Iron increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (6)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Nervous system disorders) | 0 (0) | 1 (4)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (11)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 0 (0) | 2 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 7 (8)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (4)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 10 (31)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (10)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less